CLINICAL TRIAL: NCT00222859
Title: Reasons for Nontreatment of Hepatitis C in HCV Mono-infected Patients Versus HCV-HIV Co-infected Patients in a University Setting
Brief Title: Reasons for Non-treatment of Hepatitis C in HCV Mono-infected Patients Versus HCV-HIV Co-infected Patients in a University Setting
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: IRB # 0503113
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections
Keywords: HIV; HCV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The specific aims of this study are to determine the treatment prescription rates for Hepatitis C virus (HCV) infection in a cohort of HCV mono-infected, and human immunodeficiency virus (HIV)-HCV co-infected patients and to identify the reasons for non-treatment of HCV in these two groups.

DETAILED DESCRIPTION:
Despite recent advances in treatment modalities, a large proportion of patients with HCV do not receive treatment. The reasons for non-treatment need to be elucidated to properly address these factors. Appropriate evaluation and treatment of HCV is important in providing the optimal care to these persons. It is also important to document and characterize treatment patterns and prescription rates for policy, resource allocation and funding purposes. This study will determine the rates of treatment for HCV monoinfected and HCV-HIV co-infected patients, and determine the reasons for non-treatment. It will also directly compare the two populations to determine if any differences exist in the reasons for non-treatment. This study has implications for patient care, their health outcomes, policy making, funding and resource allocation.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited from the Pittsburgh AIDS Center for Treatment (PACT) Clinic and Pitt Treatment and Evaluation Unit (PTEU) and the Center for Liver Diseases (CLD) at the University of Pittsburgh. There are approximately 800 patients in the University of Pittsburgh's PACT/PTEU clinic. Consecutive patients with HCV-HIV co-infection who present to the clinic upon initiation of data gathering would be eligible for participation in this study. An estimated 500-800 patients are seen at the CLD clinic per year, and consecutive patients enrolled in the CLD HCV registry would be considered eligible for this study. To maintain uniformity and consistency of data, only patients seen by one of the study investigators would be enrolled. Recruitment would continue till the study has enrolled 100 HCV-HIV coinfected and 200 HCV mono-infected subjects.

Exclusion Criteria:

* There are no exclusion criteria, except if the patient refuses to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HCV diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
dead or alive at end of project | December 2011

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Butt, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States